CLINICAL TRIAL: NCT05211245
Title: Comparative Evaluation of Continuous and Pulse Mode of Ultrasound Therapy in Myalgia of Maxillofacial Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr.Bhawna Saini
Record Dates: First submitted 2021-08-12; First posted 2022-01-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Myalgia; Trigger Point
Keywords: Therapeutic ultrasound
MeSH Terms: conditions — Myalgia | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse mode (Experimental): Pulsed mode of US results in nonthermal effect i.e., micro massage like which lead to segmental analgesia due to decreased central & peripheral sensitization. The non-thermal effect of US can be explain by frequency resonance theory which states that the proteins in these structures absorbs mechanical energy thus altering the structure & function, finally resulting in stimulation of phagocytosis, increase number of free radicals, increase cell membrane permeability, cellular proliferation &acceleration of fibrinolysis
  Interventions: Device: therapeutic ultrasound
- Continous mode (Active Comparator): Thermal effect which is a result of continuous mode of US therapy causes transient increase in the flexibility of collagenous structures including ligaments, tendons & joint capsules, thus leading to decrease in the pain & muscle spasm, stiffness of the joint & temporary increase in the blood flow.
  Interventions: Device: therapeutic ultrasound

INTERVENTIONS:
Device: therapeutic ultrasound — Therapeutic ultrasound ranges from 750,000 to 3,300,000 Hz (0.75 to 3.3 MHz). Depending upon the output parameters it may produce effects like increase tissue extensibility, reduction of calcium deposits, reduction of pain & muscle spasm by altering nerve conduction velocity & changes in cell membrane permeability along with increased rate of tissue repair & wound healing.There are two main types of ultrasound therapy: thermal and mechanical. Thermal effect which is a result of continuous mode of US therapy causes transient increase in the flexibility of collagenous structures including ligaments, tendons & joint capsules, thus leading to decrease in the pain & muscle spasm, stiffness of the joint & temporary increase in the blood flow. Pulsed mode of US results in nonthermal effect i.e., micro massage like which lead to segmental analgesia due to decreased central & peripheral sensitization.

SUMMARY:
Pain and trismus caused by Myalgia in masticatory muscles are one of the prime concerns for the patients. Various studies have been performed using US therapy for myofascial pain syndrome of head & neck region. US is a non-invasive frequently used physical agent which increase blood flow in tissues and collagen fibers ability to grow, & reduce muscle spasm with its thermal effect. It is difficult to imply the results of studies performed in muscles of other regions of body to the maxillofacial region because of the superficial placement of these muscles.US is being frequently used for myofascial pain, but there is an absence of a consensus regarding the frequency and mode of administration available in literature for administration of this therapy in maxillofacial region. Therefore, the present study has been designed to compare the therapeutic effect of two modes of US i.e., continuous and pulsed at 3 MHz frequency

DETAILED DESCRIPTION:
Pain and trismus caused by Myalgia in masticatory muscles are one of the prime concerns for the patients. There are limited number of studies in the literature that have evaluated therapeutic ultrasound for the management of Myalgia of maxillofacial region. Various studies have been performed, evaluating the treatment of myofascial pain with trigger point in other parts of body including neck region using ultrasound, but not all patient of myalgia present with trigger point. The most frequently used ultrasound frequencies are 1 and 3MHz. 1 MHz has more penetrating power as compared to 3MHz. Masticatory muscles being superficial in location need less penetrating waves as compared to other muscles. The ultrasound can be applied in a continuous or pulsed manner. There are studies supporting the fact that Continuous ultrasound therapy is more efficient in reducing myofascial pain syndrome of trapezius muscle at rest because it produces a heating effect in the muscles, that help in breaking the spasm. On the other hand, the pulsed mode, produces more of penetrating effect and acts on the gas bubbles of the soft tissues, thereby decreasing the inflammation. However, the two methods have not yet been compared in maxillofacial muscles. Therefore, this study aims to compare the outcome of therapeutic Ultrasound administered at 3MHz frequency in continuous & pulse modes in myalgia of maxillofacial region

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with myalgia within orofacial muscle as per DC/TMD (Ia and Ib)
2. Patient's consent for participation in this study.

Exclusion Criteria:

1. Patients with epilepsy/seizures
2. Patients with radiographic changes suggestive of pathological conditions of temporomandibular joint (TMJ).
3. Patients with undiagnosed orofacial pain
4. Any sort of skin lesion at the site where electrode is to be placed.
5. Therapeutic ultrasound must not be applied over areas of impaired circulation, ischemic areas, or areas having sensory deficit.
6. Sites of active infection
7. Patients with metal prosthesis
8. Patients with Becks depression score >25 will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the intensity of pain in each group | Base line
  Visual Analog Scale (VAS) 0n a scale of 0-10
To evaluate the intensity of pain in each group | 2 weeks
  Visual Analog Scale (VAS) 0n a scale of 0-10
To evaluate the intensity of pain in each group | 4weeks
  Visual Analog Scale (VAS) 0n a scale of 0-10
To evaluate the intensity of pain in each group | 6 weeks
  Visual Analog Scale (VAS) 0n a scale of 0-10
To evaluate the intensity of pain in each group | 3 months
  Visual Analog Scale (VAS) 0n a scale of 0-10
To assess pressure pain sensitivity of muscles in the two groups. | Base line
  Algometer
To assess pressure pain sensitivity of muscles in the two groups. | 2 weeks
  Algometer
To assess pressure pain sensitivity of muscles in the two groups. | 4 weeks
  Algometer
To assess pressure pain sensitivity of muscles in the two groups. | 6 weeks
  Algometer
To assess pressure pain sensitivity of muscles in the two groups. | 3 months
  Algometer

SECONDARY OUTCOMES:
To evaluate the maximal mouth opening and functional movements | Base line
  Digital Vernier calliper
To evaluate the maximal mouth opening and functional movements | 2 weeks
  Digital Vernier calliper
To evaluate the maximal mouth opening and functional movements | Base line ,2 weeks,4 weeks ,6 weeks, 3 months post treatment
  Digital Vernier calliper
To evaluate patient psychological status | Base line ,2 weeks,4 weeks ,6 weeks, 3 months post treatment
  Beck depression inventory
To evaluate quality of life | Base line ,2 weeks,4 weeks ,6 weeks, 3 months post treatment
  Oral Health Impact Profile (OHIP 14)
To assess the need for pain medication | Base line ,2 weeks,4 weeks ,6 weeks, 3 months post treatment
  number of medication needed

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ambika Gupta, MDS, Study Director — oral medicine & radiology,PGIDS
Locations (1):
- PGIDS, Rohtak, Haryana, India

REFERENCES:
- [Derived] Saini B, Gupta A, Singh H, Bisla S, Nagarajan S, Kumia K. Effectiveness of continuous and pulse mode of ultrasound therapy in temporomandibular disorders associated myalgia-a randomized controlled study. J Oral Facial Pain Headache. 2025 Mar;39(1):81-92. doi: 10.22514/jofph.2025.007. Epub 2025 Mar 12. PMID 40129425